CLINICAL TRIAL: NCT07013604
Title: Effectiveness of Neuromuscular Electrical Stimulation Versus Low-load Resistance Training With Blood Flow Restriction in Elderly Individuals With Sarcopenia
Brief Title: Sarcopenia and Intervention Physical Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, Ola Mohamed Elsayed Elgohary, ola mohamed elsayed elgohary, Pharos University in Alexandria
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: sarcopenia
Record Dates: First submitted 2025-05-29; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: This study follows a randomised controlled trial (RCT) design involving 60 elderly participants aged 60-75 years diagnosed with sarcopenia according to EWGSOP2 criteria. Participants will be randomly assigned to three groups (n = 20 each).
Who Masked: Participant
Masking Description: This study uses single-blind masking. While participants are aware of their group assignment due to the nature of the interventions (especially NMES and resistance training), outcome assessors who perform the post-intervention evaluations (e.g., muscle strength, functional performance, and quality of life) will be blinded to group allocation. This is done to reduce assessment bias and ensure objective measurement of outcomes.
  Additionally, the control group receives a placebo treatment (being connected to a non-active neuromusculoskeletal device), which helps reduce the psychological effects of knowing they are not receiving active intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neuromuscular Electrical Stimulation (NMES) Group (Experimental): Participants receive neuromuscular electrical stimulation (NMES) targeting the quadriceps and hamstrings, 30 minutes per session, 3 times per week for 8 weeks
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES) Group,Resistance + BFR Group
- Resistance + BFR Group (Experimental): Participants perform low-load resistance training (30% 1RM) combined with blood flow restriction using pneumatic cuffs, 30 minutes per session, 3 times per week for 8 weeks
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES) Group,Resistance + BFR Group
- Control Group (Placebo Comparator): Participants receive placebo treatment by being connected to a neuromusculoskeletal device that is turned off (no actual stimulation), with no active intervention during the 8-week period
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES) Group,Resistance + BFR Group

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation (NMES) Group,Resistance + BFR Group — NMES Group: Receives neuromuscular electrical stimulation to the thigh muscles for 30 minutes, three times per week, over 8 weeks.
  Resistance + BFR Group: Performs low-load resistance exercises with blood flow restriction applied to the thighs, also for 30 minutes per session, three times per week, over 8 weeks.
  Control Group: Receives placebo treatment using a turned-off stimulation device with no active intervention during the 8-week period.

SUMMARY:
To evaluate and compare the effectiveness of neuromuscular electrical stimulation (NMES) and low-load resistance training with blood flow restriction (BFR) in improving muscle mass, strength, functional performance, and quality of life in elderly individuals diagnosed with sarcopenia

DETAILED DESCRIPTION:
Sarcopenia, the age-related decline in muscle mass, strength, and function, significantly affects the health and independence of elderly individuals. It increases the risk of frailty, falls, and disability. Neuromuscular electrical stimulation (NMES) and low-load resistance training with blood flow restriction (BFR) are promising rehabilitation strategies for older adults with limited physical capacity. This study aims to compare the effectiveness of NMES and BFR in managing sarcopenia and improving physical and functional outcomes in the elderly

ELIGIBILITY:
Inclusion Criteria:

* Older age (≥ 60-75 years)

Low muscle strength (e.g., low handgrip strength)

Low muscle mass (e.g., ASM/height² below cutoff)

Exclusion Criteria:

* heart disese
* kidny disese
* autoimune disese
* cognetive disorder
* sever form of sarcopenia

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle Mass | 2 month
  Assessed using Bioelectrical Impedance Analysis (BIA) to measure skeletal muscle mass.
  Evaluation is done pre- and post-intervention to detect changes in the Skeletal Muscle Index (SMI), based on EWGSOP2 criteria

SECONDARY OUTCOMES:
Muscle Strength Handheld dynamometer (e.g., MicroFET) | 2 month
  Isometric knee extension strength
  Measurement: Pre- and post-intervention, using the highest or average value from 2-3 trials.
Timed Up and Go (TUG) Test | 2 month
  Assesses eight domains of health-related quality of life, scored from 0 to 100. Administered before and after the intervention period